CLINICAL TRIAL: NCT03323008
Title: E-training of Inmate Peer Caregivers for Enhancing Geriatric and End-of-life Care in Prisons
Acronym: P2P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); Penn State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1R41AG057239-01 (NIH); 1R41AG057239-01 (NIH); 03017 (Other: Klein Buendel, Inc.)
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Aging Problems
Keywords: Prisoners; End-of-life Care; Geriatric Care; Palliative Care; Hospice Care; Prison; Corrections; Inmates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training Prototype (Experimental): Testing of 3 modules
  Interventions: Other: Prototype

INTERVENTIONS:
Other: Prototype — Usability testing and System Usability Scale

SUMMARY:
The mission of corrections is to provide care, custody, and control for incarcerated individuals. United State prisons are required by constitutional law to provide adequate care for growing numbers of older inmates who will likely spend their final days in prison. This Phase I project focuses on research and development of highly interactive computer-based learning modules for inmate peer caregivers to promote an integrated systems approach to enhancing the care of the aged and dying in prisons.

DETAILED DESCRIPTION:
The US has the highest incarceration rate in the world-imprisoning 693 people per 100,000. The older adult segment of the prison population has more than tripled since 1990 and their health issues are common to free people who are 10-15 years their senior. Inmates over the age of 55 have a death rate that is 10 times that of prisoners aged 25-34. US prison systems are facing sharply increased demands in caring for aged and dying inmates. A recent systematic review revealed that inmate peer caregivers can figure prominently in delivery of end-of-life (EOL) care in prison. However, the degree of training received by inmate peer caregivers varies widely. The lack of consistent training, both in content and duration points to a need for evidence based, current, and readily accessible training for this abundant human resource for meeting a growing need in US prisons. In response to this need, this Phase I STTR project, titled E-training of Inmate Peer Caregivers for Enhancing Geriatric and End-of-Life Care in Prisons, will demonstrate the scientific merit and feasibility of developing cutting edge, media rich learning modules to train inmate peer caregivers in geriatric and EOL care. The specific aims of the project are to (1) transform best practices in inmate peer caregiving into a comprehensive training program that consists of media-rich and highly interactive computer-based learning modules for providing geriatric and EOL care to their peers; and (2) conduct in-person usability testing of the media-rich and highly interactive web-based prototypes with inmates who are currently Mental Health Peer Support Specialists (i.e., prisoners who are experienced caregivers, but naïve to geriatric and EOL care) to evaluate the user interface, ease of use, and perceived barriers in order to refine and optimize the product. In collaboration with an advisory board of experts in prison healthcare, geriatrics, ethics, palliative/hospice care, and oversight of an inmate peer support program, the investigators plan and develop discussion guides and then conduct focus groups with three groups of prison stakeholders: inmates who serve as peer caregivers for aged or dying peers; interdisciplinary staff who care for, or oversee care of aged and dying inmates; and training and information technology staff. One focus group with each of the above three constituent groups will be held at a men's and a women's prison. Focus groups will permit investigators to ensure that the design and technology plans match what is allowable for inmate training and will allow us to isolate essential geriatric and EOL content for specification in the development of the comprehensive training program. Finally, the investigators will create and evaluate prototypes of media rich, interactive computer-based learning modules for inmates serving as peer caregivers. At the end of Phase I, the investigators will have a specifications document for the design of modules that: fit with the technology available in corrections settings; is permissible to be used by inmates; represents the critical learning needs of inmate peer caregivers for assisting with geriatric and EOL care; and further develops the collaborative relationships in preparation for commercialization of the product.

ELIGIBILITY:
Inmate Inclusion Criteria:

* Be a Mental Health Peer Support Specialist
* Be 18 years or older
* Able to speak, understand, and read English
* Able to consent.

Inmate Exclusion Criteria:

* Not be a Mental Health Peer Support Specialist
* Under 18 years of age
* Unable to speak, understand, and read English
* Unable to consent.

Prison Employee Inclusion Criteria:

* 18 years or older
* Employed by a participating at a participating prison
* Able to speak, understand, and read English
* Able to consent

Prison Employee Exclusion Criteria:

* Under 18 years
* Not employed by a participating prison
* Unable to speak English
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
System Usability Scale | 2 months
  The System Usability Scale (SUS) is a validated tool for assessing the usability and acceptability of technology-based products. It contains 10 questions that are rated on a scale from 1 to 5. "The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100." A score of 68 is considered "above average." Anything below a 68 is considered "below average." The higher the score, the higher the usability of the product.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Myers, PHD, Principal Investigator — Klein Buendel, Inc.
Locations (2):
- United States (2):
  - Klein Buendel, Inc., Golden, Colorado
  - Penn State University, University Park, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loeb SJ, Steffensmeier D, Lawrence F. Comparing incarcerated and community-dwelling older men's health. West J Nurs Res. 2008 Mar;30(2):234-49; discussion 250-8. doi: 10.1177/0193945907302981. Epub 2007 Jul 13. PMID 17630382
- [Background] Noonan M, Ginder S. Mortality in local jails and state prisons, 2000-2012-statistical table. Washington, DC: US Department of Justice, Office of Justice Programs, Bureau of Justice Statistics. October 2014.
- [Background] Wion RK, Loeb SJ. CE: Original Research: End-of-Life Care Behind Bars: A Systematic Review. Am J Nurs. 2016 Mar;116(3):24-36; quiz 37. doi: 10.1097/01.NAJ.0000481277.99686.82. PMID 26871892
- [Background] Cloyes KG, Rosenkranz SJ, Berry PH, Supiano KP, Routt M, Shannon-Dorcy K, Llanque SM. Essential Elements of an Effective Prison Hospice Program. Am J Hosp Palliat Care. 2016 May;33(4):390-402. doi: 10.1177/1049909115574491. Epub 2015 Mar 2. PMID 25735806